CLINICAL TRIAL: NCT03301077
Title: The Mental Health in Austrian Teenagers (MHAT) - Study: First Epidemiological Survey
Brief Title: Mental Health in Austrian Teenagers (MHAT)
Acronym: MHAT
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Ludwig Boltzmann Institut Health Promotion Research (Unknown); Pharmig - Gesundheitsziele aus dem Rahmen-Pharmavertrag (Other)
Responsible Party: Principal Investigator, Dr. Andreas Karwautz, Univ. Prof. Dr., Medical University of Vienna
Other Study IDs: FA765A0303
Record Dates: First submitted 2014-07-21; First posted 2017-10-04 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Mental Disorders
Keywords: children and adolescents; mental health; epidemiology; psychiatric disorders
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being | interventions — Mass Screening; Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- General population: recruited from schools and other institutions like job-centers or child and adolescent psychiatries
  Interventions: Other: 2-phase epidemiological study (screening, interviews)

INTERVENTIONS:
Other: 2-phase epidemiological study (screening, interviews) — first phase is the screening phase, second phase is the interview phase

SUMMARY:
The purpose of the Mental Health in Austrian Teenagers (MHAT) - Study is to collect the first epidemiological data on mental health and psychiatric disorders in a representative sample of Austrian adolescents between 10 and 18 years.

DETAILED DESCRIPTION:
Knowing about the prevalence of psychiatric disorders and related risk and protective factors is essential for the development of prevention programs and therapeutic approaches. Up to now, no epidemiological data on prevalence rates of psychiatric disorders and related risk and protective factors based on a representative sample is available for Austrian adolescents.

The aim of the study is to present rates of behavioral, emotional and social problems as well as prevalence rates of mental disorders. Furthermore the investigators want to examine risk factors, protective factors and quality of life in a large sample of adolescents aged 10 to 18 years. A two step design is chosen for this purpose to obtain diagnoses based on the Diagnostic and Statistical Manual of the American Psychiatric Association, Version 5 (DSM-5):

1. Phase 1 (screening) is a screening for emotional, behavioral and social problems as well as social and demographic correlates, risk and protective factors and quality of life.
2. Phase 2 (interviews) includes structured diagnostic interviews to assess psychiatric diagnoses according to DSM-5 criteria with adolescents above a predefined cut-off score in the screening, and a random sample of adolescents scoring below the cut-off.

ELIGIBILITY:
Inclusion Criteria:

* adolescents aged 10-18

Exclusion Criteria:

* no written informed consent possible due to intelligence or no willingness by parents to include minor

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: general population
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2013-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
psychiatric problems (diagnoses based on the Diagnostic and Statistical Manual of the American Psychiatric Association, Version 5 (DSM-5) | 12 months
  Screening and interview

SECONDARY OUTCOMES:
rates of behavioral, emotional and social problems (representation of data collected at interview) | 12 months
  YSR (Youth Self Report) questionnaire
psychiatric disorder related risks and protective factors (representation of data collected at interviews) | 12 months
  Kinder-DIPS (Diagnostisches Interview psychischer Störungen) interview
quality of life (total score, self-perception, parent relation & home life, social support & peers, school environment and bullying) | 12 months
  KIDSCREEN (Kidscreen) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Karwautz, MD, Prof, Study Director — Medical University Vienna; Wolfgang Dür, Phd, Prof, Study Director — Ludwig Boltzmann Institute LBIHPR
Locations (1):
- Medical University of Vienna, Dep. of Child and Adolescent Psychiatry, Vienna, Austria

REFERENCES:
- See also: Related Info — http://www.ess-stoerung.eu